CLINICAL TRIAL: NCT06907498
Title: Paromomycin or Metronidazole for Symptomatic Dientamoeba Fragilis in Adults (COMFORTER Trial) - Protocol for a Superiority Double Blind, Randomized Controlled Trial
Brief Title: Paromomycin or Metronidazole for Symptomatic Dientamoeba Fragilis in Adults
Acronym: COMFORTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Dafna Yahav, Head, Infectious Diseases Unit, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D. fragilis treatment
Record Dates: First submitted 2023-12-20; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Dientamoeba Fragilis Infection
Keywords: Dientamoeba Fragilis; Diarrhea; Paromomycin; Metronidazole; Treatment
MeSH Terms: conditions — Dientamoebiasis; Diarrhea | interventions — Paromomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paromomycin (Experimental): Paromomycin 500mg X3 / day
  Interventions: Drug: Paromomycin
- Metronidazole (Active Comparator): Metronidazole 500mg X3 / day
  Interventions: Drug: Paromomycin

INTERVENTIONS:
Drug: Paromomycin — Paromomycin 500mg X3 / day
  Other Names: Kaman

SUMMARY:
Dientameba Fragilis (D.fragilis) is a protozoan found in the digestive tract - in the human colon. there are disagreements regarding the preferred treatment for these cases, with several regimens tested in mostly small observational studies. Several drugs are currently recommended for D.fragilis, with metronidazole most commonly used. However, metronidazole therapy for treating dientamoebiasis in children was not associated with better clinical outcomes in a randomized, double-blinded and placebo-controlled clinical trial.

Hence, we aim to perform a double blind, randomized controlled trial, evaluating the clinical and microbiological efficacy of paromomycin versus metronidazole for the treatment of symptomatic adults with PCR positive dientamoeba fragilis.

The primary outcomes would be clinical improvement or resolution. Secondary outcomes include clinical improvement evaluated by a visual analogue scale; microbiological eradication, quality of life, and adverse events related to therapy.

We plan to include 60 patients (30 per arm)

DETAILED DESCRIPTION:
Introduction Dientameba Fragilis (D.fragilis) is a protozoan found in the digestive tract - in the human colon. The route of transmission is fecal-oral, and infection can lead to chronic gastrointestinal symptoms manifested by abdominal pain, diarrhea, abdominal bloating, anal pruritus, and in addition pronounced fatigue [1]. Since the introduction of a molecular diagnosis [PCR] for a stool test, it has become clear that these protozoa are a main protozoa inhabiting the digestive system, with stool positivity rates ranging from 12 to 68%, depending on country and age [2].

This parasite was first identified about 100 years ago and since then debates have continued in the medical literature as to whether it is indeed a pathogen or a commensal [3]. In addition, there are disagreements regarding the preferred treatment for these cases, with several regimens tested in mostly small observational studies. Several drugs are currently recommended for D.fragilis, with metronidazole most commonly used [4]. However, metronidazole therapy for treating dientamoebiasis in children was not associated with better clinical outcomes in a randomized, double-blinded and placebo-controlled clinical trial. Furthermore despite observing higher eradication rates two weeks after end of therapy with metronidazole in this trial, positivity rebounded quickly appeared after therapy. [5]. In contrast, several observational studies have reported high clinical and microbiological success rates with paromomycin, with over 80% eradication in adults [6,7]. We could not identify any prospective study comparing head to head these two drugs; metronidazole and paromomycin.

In light of the above, we plan to perform a double blind, randomized controlled trial, evaluating the clinical and microbiological efficacy of paromomycin versus metronidazole for the treatment of symptomatic adults with PCR positive dientamoeba fragilis.

The primary outcomes is clinical improvement or resolution (yes/no. Secondary outcomes include clinical improvement evaluated by a visual analogue scale; microbiological eradication, quality of life, and adverse events related to therapy.

Aim

* To evaluate clinical response to paromomycin versus metronidazole treatment.
* To evaluate whether paromomycin is superior to metronidazole in eradicating D. fragilis in molecular stool testing (PCR) 3-4 weeks after end of therapy.
* Additional aim is to evaluate the relationship between clinical cure and eradication of the parasite.

Design: Double-blind Randomized Controlled study comparing metronidazole vs. paromomycin treatment in patients with prolonged gastrointestinal symptoms and positive D. fragilis in molecular (PCR) stool test.

Patients will be approached through social networks advertisements, infectious diseases and gastrointestinal clinics, inviting individuals suffering from gastrointestinal symptoms over one month who had a positive PCR test for D. fragilis in the previous 6 months. These patients will be invited for a clinic visit.

Population:

Inclusion criteria: Patients over the age of 18, not including pregnant women - With persistent gastrointestinal symptoms (over one month).

* Without any other clear diagnosis to explain these symptoms according to medical records.
* With a positive PCR stool test for D. fragilis without any additional pathogen (patients with Blastocystis hominis in feces will not be excluded).

Exclusion criteria:

* Pregnancy
* Hypersensitivity to any of the study drugs or to aminoglycosides
* Patients age below 18 years
* Metronidazole or paromomycin treatment in the last 3 months

Intervention: After signing informed consent, study participants will fill out symptoms questionnaire, built in 4-point Likert scale (See Appendix).

We will randomize them into two treatment arms: paromomycin and metronidazole. Randomization will be generated by computer and will be central. Study allocation will be blinded from patients, principal investigators and outcome assessors.

Medical treatment planned for 7 days as follows:

1. Metronidazole 500mg X3 / day
2. Paromomycin 500mg X3 / day In both preparations the pill is 250 mg, so both treatment arms will have the same number of tabs and same length of treatment. Patients will be provided with the drugs for 7 days (we will examine the possibility of making it identical in appearance).

Follow-up

1. Monitoring side effects for each drug - using a questionnaire. This will be conducted by telephone at the end of the treatment (one week) by a research assistant (without passing the information to the doctor - to prevent revealing of blinding).
2. In person meeting with a study physician 3-4 weeks after completion of treatment, at which time the patient will fill out a structured questionnaire for symptom evaluation (See Appendix). The physician will be blinded to the patient's treatment. Clinical improvement will be defined as improvement in the Likert scale in at least one symptom, with no exacerbation in any other symptom.
3. Repeated PCR stool test 3-4 weeks after the end of treatment.
4. An additional similar visit will be held at 8 and 12 weeks after end to treatment.

Sample size calculation for superiority:

In order to show superiority of paromomycin with 90% power and an Alpha of 5%, assuming 80% clinical improvement with paromomycin versus 40% with metronidazole, a sample size of 27 patients per arm will be required. Considering a dropout rate of up to 10%, we estimate a sample size of 60 patients.

ELIGIBILITY:
Inclusion Criteria:

Patients over the age of 18, not including pregnant women - With persistent gastrointestinal symptoms (over one month).

* Without any other clear diagnosis to explain these symptoms according to medical records.
* With a positive PCR stool test for D. fragilis without any additional pathogen (patients with Blastocystis hominis in feces will not be excluded).

Exclusion Criteria:

* Pregnancy
* Hypersensitivity to any of the study drugs or to aminoglycosides
* Patients age below 18 years
* Metronidazole or paromomycin treatment in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
clinical improvement or resolution | 30 day
  clinical improvement or resolution

SECONDARY OUTCOMES:
clinical improvement by a visual analogue scale | 30 day
  clinical improvement by a visual analogue scale
microbiological eradication | 30 day
  microbiological eradication - negative PCR
Quality of life scale | 30 day
  Quality of life scale
Adverse events | 30 day
  Adverse events - gastrointestinal, neurological

CONTACTS AND LOCATIONS:
Overall Officials: Dafna Yahav, MD, Principal Investigator — Sheba Medical Center, Ramat-Gan, Israel
Locations (1):
- Sheba medical center, Ramat Gan, Israel, Israel

IPD SHARING:
Plan to Share IPD: Yes
IPD would be shared in case of reasonable request from the PI
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Within 90 days from study completion and for 1 year
Access Criteria: By request from PI